CLINICAL TRIAL: NCT00093795
Title: A Phase III, Adjuvant Trial Comparing Three Chemotherapy Regimens in Women With Node-Positive Breast Cancer: Docetaxel/Doxorubicin/Cyclophosphamide (TAC); Dose-Dense (DD) Doxorubicin/Cyclophosphamide Followed By DD Paclitaxel (DD AC→P); DD AC Followed By DD Paclitaxel Plus Gemcitabine (DD AC→PG)
Brief Title: Combination Chemotherapy in Treating Women Who Have Undergone Surgery for Node-Positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-38; U10CA012027 (NIH); NCT00191958 (obsolete NCT alias)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Gemcitabine; Paclitaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: TAC X 6 (Active Comparator): Doxorubicin, cyclophosphamide, and docetaxel.
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin
- Group 2: AC X 4 then P X 4 (Active Comparator): Doxorubicin, cyclophosphamide, and paclitaxel
  Interventions: Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Doxorubicin
- Group 3: AC X 4 then PG X 4 (Experimental): Doxorubicin, cyclophosphamide, paclitaxel and gemcitabine
  Interventions: Drug: Cyclophosphamide; Drug: Gemcitabine; Drug: Paclitaxel; Drug: Doxorubicin

INTERVENTIONS:
Drug: Cyclophosphamide — Group 1: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
  Group 2 and Group 3: cyclophosphamide 600 mg/m2 IV every 14 days for 4 cycles
  Other Names: C
Drug: Docetaxel — 75 mg/m2 IV every 21 days for 6 cycles
  Other Names: Taxotere; T
  Arms: Group 1: TAC X 6
Drug: Gemcitabine — 2000 mg/m2 IV every 14 days for 4 cycles
  Other Names: Gemzar; G
  Arms: Group 3: AC X 4 then PG X 4
Drug: Paclitaxel — 175 mg/m2 IV every 14 days for 4 cycles
  Other Names: Taxol; P
  Arms: Group 2: AC X 4 then P X 4; Group 3: AC X 4 then PG X 4
Drug: Doxorubicin — Group 1: 50 mg/m2 IV every 21 days for 6 cycles
  Group 2 and Group 3: 60 mg/m2 IV every 14 days for 4 cycles
  Other Names: A; Adriamycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, doxorubicin , cyclophosphamide, paclitaxel, and gemcitabine work in different ways to stop tumor cells from dividing so they stop growing or die. Giving combination chemotherapy after surgery may kill any remaining tumor cells.

PURPOSE: This randomized phase III trial is studying three different combination chemotherapy regimens and comparing how well they work in treating women who have undergone surgery for node-positive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare disease-free survival in women with node-positive breast cancer treated with 3 different adjuvant chemotherapy regimens comprising dose-dense doxorubicin, cyclophosphamide, paclitaxel, and gemcitabine vs docetaxel, doxorubicin, and cyclophosphamide vs dose-dense doxorubicin, cyclophosphamide, and paclitaxel.

Secondary

* Compare overall survival, recurrence-free interval, and distant recurrence-free interval, in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to number of positive lymph nodes (1-3 vs 4-9 vs ≥ 10), hormone receptor status (estrogen receptor [ER]- and progesterone receptor [PgR]- negative vs ER- and/or PgR-positive), type of prior surgery and planned radiotherapy (lumpectomy and local radiotherapy [RT] without regional RT vs lumpectomy and local RT with regional RT vs mastectomy without RT vs mastectomy with local or regional RT). Patients are randomized to 1 of 3 treatment arms.

* Group 1: Patients receive doxorubicin IV over 15 minutes, cyclophosphamide IV over 30 minutes, and docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for 6 courses.
* Group 2: Patients receive AC chemotherapy comprising doxorubicin IV over 15 minutes and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 14 days for 4 courses. Beginning 14 days after the last dose of AC, patients receive paclitaxel IV over 3 hours on day 1. Treatment repeats every 14 days for 4 courses.
* Group 3: Patients receive AC chemotherapy as in Group 2. Beginning 14 days after the last dose of AC, patients receive paclitaxel as in Group 2 and gemcitabine IV over 30-60 minutes on day 1. Treatment repeats every 14 days for 4 courses.

In all arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Beginning 3-12 weeks after the last dose of chemotherapy, patients with ER-positive and/or PgR-positive tumors receive hormonal therapy.

Beginning no sooner than 3 weeks after the last dose of chemotherapy, patients treated with lumpectomy undergo whole-breast radiotherapy. Patients treated with mastectomy may undergo chest wall and/or regional nodal radiotherapy.

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 4,800 patients will be accrued for this study within 4 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must consent to participate in the study and must have signed an approved consent form conforming with federal and institutional guidelines.
* The patient must have a life expectancy of at least 10 years and a Zubrod performance status of 0 or 1. (Comorbid conditions but not the diagnosis of breast cancer should be taken into consideration when determining life expectancy.)
* The interval between the last surgery for breast cancer staging or treatment and randomization must be no more than 84 days.
* The tumor must be invasive carcinoma of the breast on histologic examination.
* All of the following staging criteria must be met:

  * By clinical and pathologic evaluation, primary tumor must be T1-3;
  * By clinical evaluation, ipsilateral nodes must be cN0, cN1, or cN2a;
  * By pathologic evaluation, ipsilateral nodes must be pN1 (pN1mi, pN1a, pN1b, pN1c), pN2a, pN3a, or pN3b (only if due to microscopic involvement of internal mammary node detected by sentinel lymph node dissection and with more than 3 positive axillary lymph nodes).
* Patients must have an estrogen receptor (ER) analysis performed on the primary tumor prior to randomization. If ER analysis is negative, then progesterone receptor (PgR) analysis must be performed. If ER analysis is positive, PgR analysis is desired, but not mandatory. ("Marginal" or "borderline" results [i.e., those not definitely negative] will be considered positive regardless of the methodology used.)
* Patients must have had either a lumpectomy or a total mastectomy. Patients must have completed one of the following procedures for evaluation of pathologic nodal status.

  * Sentinel lymphadenectomy followed by removal of additional non-sentinel lymph nodes (This approach is strongly recommended.)
  * Sentinel lymphadenectomy alone if one of the following criteria is met:
  * Pathologic nodal staging based on sentinel lymphadenectomy is pN1mi or pN1b
  * Surgeon elects not to remove additional non-sentinel nodes (This approach is strongly discouraged, but will not preclude participation in B-38.)
  * Axillary lymphadenectomy without sentinel node isolation procedure.
* Patients must have no clinical or radiologic evidence of metastatic disease.
* Patients with either skeletal pain or alkaline phosphatase that is greater than ULN but less than or equal to 2.5 x ULN are eligible for inclusion in the study if bone scans fail to demonstrate metastatic disease. Suspicious findings on bone scan must be confirmed as benign by x-ray, MRI, or biopsy.
* Patients with aspartate transaminase (AST) or alkaline phosphatase greater than ULN are eligible for inclusion in the study if liver imaging fails to demonstrate metastatic disease and the following requirements are met at the time of randomization.

  * Postoperative absolute granulocyte count (AGC) must be greater than or equal to 1200/mm3.
  * Postoperative platelet count must be greater than or equal to 100,000/mm3.
  * The following criteria for postoperative evidence of adequate hepatic function must be met:

    * total bilirubin must be less than or equal to ULN for the lab unless the patient has a grade 1 bilirubin elevation (greater than ULN to 1.5 x ULN) due to Gilbert's disease or similar syndrome due to slow conjugation of bilirubin; and
    * alkaline phosphatase must be less than or equal to 2.5 x ULN for the lab; and
    * the AST must be less than or equal to 1.5 x ULN for the lab; and
    * alkaline phosphatase and AST cannot both be greater than ULN.
  * Postoperative serum creatinine must be less than or equal to ULN.
* At the time of randomization, the patient must have had the following: history and physical exam, EKG, and imaging of the chest within the past 3 months and bilateral mammogram within the past 6 months.
* Within 3 months prior to entry, the patient must have a baseline left ventricular ejection fraction (LVEF), measured by Multiple Gated Acquisition (MUGA) scan or echocardiogram, greater than or equal to lower limit of normal (LLN) for the facility performing the procedure and no evidence of regional wall abnormalities.
* Patients with a history of non-breast malignancies are eligible if they have been disease-free for 5 or more years prior to randomization and are deemed by their physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Special conditions for eligibility of lumpectomy patients: radiation therapy and surgery. Patients treated by lumpectomy must meet all the eligibility criteria in addition to the following:

  * Generally, lumpectomy should be reserved for tumors less than 5 cm. However, at the investigator's discretion, patients treated with lumpectomy for tumors greater than or equal to 5 cm are eligible if eligibility criteria for lumpectomy are met.
  * The margins of the resected specimen must be histologically free of invasive tumor and DCIS as determined by the local pathologist. In patients for whom pathologic examination demonstrates tumor present at the line of resection, additional operative procedures may be performed to obtain clear margins. This is permissible even if axillary evaluation has been completed. Patients in whom tumor is still present at the resected margin after re-excision(s) must undergo total mastectomy to be eligible. (Patients with margins positive for lobular carcinoma in situ (LCIS) are eligible without additional resection.)
  * Irradiation of regional lymph nodes is optional, but plans for radiation therapy must be declared by the investigator prior to randomization for stratification purposes.
* Special conditions for eligibility of mastectomy patients: radiation therapy o Postmastectomy chest wall and/or regional nodal irradiation is optional. Plans for radiation in mastectomy patients must be declared by the investigator prior to randomization for stratification purposes.

Ineligibility Criteria

* Male patients are not eligible for this study. Women with one or more of the following conditions or prior therapies are also ineligible for this study:
* Tumor that has been determined to be human epidermal growth factor receptor 2 (HER2)-positive by immunohistochemistry (3+) or by fluorescent in situ hybridization (positive for gene amplification).
* Contralateral breast cancer (invasive or DCIS) or a mass or mammographic abnormality in the opposite breast suspicious for malignancy unless there is biopsy proof that the mass is not malignant.
* Primary tumor staged as T4 for any reason.
* Clinical nodal stages including cN2b and cN3 or pathologic nodal stages including pN0(i+), pN2b, pN3b with clinically apparent internal mammary nodes, or pN3c.
* Suspicious nodes in the contralateral axilla or suspicious supraclavicular nodes. Patients with these conditions are considered ineligible unless there is biopsy evidence that these are not involved with tumor.
* Prior history of breast cancer, including DCIS (patients with a history of LCIS are eligible).
* Treatment, including radiation therapy, chemotherapy, and/or hormonal therapy administered for the currently diagnosed breast cancer prior to randomization. One exception is hormonal therapy, which may have been given for up to a total of 28 days anytime after diagnosis and before study entry. In such a case, hormonal therapy must stop at or before randomization and be re-started, if indicated, following chemotherapy. A second exception is radiation therapy for patients enrolled in NSABP B-39 and assigned to partial breast irradiation (Group 2). These patients may have received RT prior to B-38 study entry.
* Prior therapy with anthracyclines or taxanes for any malignancy.
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormonal replacement therapy, etc. (These patients are eligible if this therapy is discontinued prior to randomization.)
* Therapy with any hormonal agents such as raloxifene (Evista®), tamoxifen, or other selective estrogen-receptor modulators (SERMs), either for osteoporosis or breast cancer prevention. (Patients are eligible only if these medications are discontinued prior to randomization.
* Cardiac disease that would preclude the use of anthracyclines. This includes:

  * history of myocardial infarction documented by elevated cardiac enzymes or regional wall abnormalities on assessment of left ventricular (LV) function;
  * angina pectoris that requires the use of anti-anginal medication;
  * any history of documented congestive heart failure;
  * serious cardiac arrhythmia requiring medication;
  * severe conduction abnormality;
  * valvular disease with documented cardiac function compromise; and
  * uncontrolled hypertension defined as blood pressure greater than 160/100 on antihypertensive therapy.
* Conditions that would prohibit administration of corticosteroids.
* Sensory/motor neuropathy greater than or equal to grade 2, as defined by the NCI's Common Terminology Criteria for Adverse Events Version 3.0.
* Non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude a patient from receiving any of the treatment options or would prevent prolonged follow-up.
* History of hepatitis B or C.
* Pregnancy or lactation at the time of proposed randomization. Women of reproductive potential must agree to use an effective non-hormonal method of contraception.
* Concurrent treatment with other investigational agents for the treatment of breast cancer.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Special conditions for ineligibility of lumpectomy patients: radiation therapy and surgery

  * For patients treated by lumpectomy, whole breast irradiation is required.
  * The following patients will be ineligible:
  * Patients with diffuse tumors (as demonstrated on mammography) treated with lumpectomy. (These patients are eligible if they undergo mastectomy.)
  * Patients treated with lumpectomy in whom there is another clinically dominant mass or mammographically suspicious abnormality within the ipsilateral breast remnant. Such a mass must be biopsied and demonstrated to be histologically benign prior to randomization or, if malignant, must be surgically removed with clear margins.
  * Patients in whom the margins of the resected specimen are involved with invasive tumor or DCIS.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4894 (Actual)
Dates: Start 2004-10; Primary Completion 2012-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (12):
- United States (12):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - Robert and Carol Weissman Cancer Center at Martin Memorial, Stuart, Florida
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - South Shore Hospital, South Weymouth, Massachusetts
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Chestnut Hill Healthcare Cancer Center, Philadelphia, Pennsylvania
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington

REFERENCES:
- [Derived] Swain SM, Tang G, Geyer CE Jr, Rastogi P, Atkins JN, Donnellan PP, Fehrenbacher L, Azar CA, Robidoux A, Polikoff JA, Brufsky AM, Biggs DD, Levine EA, Zapas JL, Provencher L, Northfelt DW, Paik S, Costantino JP, Mamounas EP, Wolmark N. Definitive results of a phase III adjuvant trial comparing three chemotherapy regimens in women with operable, node-positive breast cancer: the NSABP B-38 trial. J Clin Oncol. 2013 Sep 10;31(26):3197-204. doi: 10.1200/JCO.2012.48.1275. Epub 2013 Aug 12. PMID 23940225

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: TAC X 6: Doxorubicin, cyclophosphamide, and docetaxel.
  Cyclophosphamide: Group 1: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
  Group 2 and Group 3: cyclophosphamide 600 mg/m2 IV every 14 days for 4 cycles
  Docetaxel: 75 mg/m2 IV every 21 days for 6 cycles
  Doxorubicin: Group 1: 50 mg/m2 IV every 21 days for 6 cycles
  Group 2 and Group 3: 60 mg/m2 IV every 14 days for 4 cycles
- Group 2: AC X 4 Then P X 4: Doxorubicin, cyclophosphamide, and paclitaxel
  Cyclophosphamide: Group 1: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
  Group 2 and Group 3: cyclophosphamide 600 mg/m2 IV every 14 days for 4 cycles
  Paclitaxel: 175 mg/m2 IV every 14 days for 4 cycles
  Doxorubicin: Group 1: 50 mg/m2 IV every 21 days for 6 cycles
  Group 2 and Group 3: 60 mg/m2 IV every 14 days for 4 cycles
- Group 3: AC X 4 Then PG X 4: Doxorubicin, cyclophosphamide, paclitaxel and gemcitabine
  Cyclophosphamide: Group 1: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
  Group 2 and Group 3: cyclophosphamide 600 mg/m2 IV every 14 days for 4 cycles
  Gemcitabine: 2000 mg/m2 IV every 14 days for 4 cycles
  Paclitaxel: 175 mg/m2 IV every 14 days for 4 cycles
  Doxorubicin: Group 1: 50 mg/m2 IV every 21 days for 6 cycles
  Group 2 and Group 3: 60 mg/m2 IV every 14 days for 4 cycles
Period: Overall Study
Arm/Group | Group 1: TAC X 6 | Group 2: AC X 4 Then P X 4 | Group 3: AC X 4 Then PG X 4
Started | 1630 | 1634 | 1630
Completed | 1610 | 1618 | 1613
Not Completed | 20 | 16 | 17
Not completed — No follow up data | 20 | 16 | 17

BASELINE CHARACTERISTICS:
Groups:
- TAC X 6: Doxorubicin, cyclophosphamide, and docetaxel. Cyclophosphamide: Group 1: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles Group 2 and Group 3: cyclophosphamide 600 mg/m2 IV every 14 days for 4 cycles Docetaxel: 75 mg/m2 IV every 21 days for 6 cycles Doxorubicin: Group 1: 50 mg/m2 IV every 21 days for 6 cycles Group 2 and Group 3: 60 mg/m2 IV every 14 days for 4 cycles
- AC X 4 Then P X 4: Doxorubicin, cyclophosphamide, and paclitaxel Cyclophosphamide: Group 1: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles Group 2 and Group 3: cyclophosphamide 600 mg/m2 IV every 14 days for 4 cycles Paclitaxel: 175 mg/m2 IV every 14 days for 4 cycles Doxorubicin: Group 1: 50 mg/m2 IV every 21 days for 6 cycles Group 2 and Group 3: 60 mg/m2 IV every 14 days for 4 cycles
- AC X 4 Then PG X 4: Doxorubicin, cyclophosphamide, paclitaxel and gemcitabine Cyclophosphamide: Group 1: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles Group 2 and Group 3: cyclophosphamide 600 mg/m2 IV every 14 days for 4 cycles Gemcitabine: 2000 mg/m2 IV every 14 days for 4 cycles Paclitaxel: 175 mg/m2 IV every 14 days for 4 cycles Doxorubicin: Group 1: 50 mg/m2 IV every 21 days for 6 cycles Group 2 and Group 3: 60 mg/m2 IV every 14 days for 4 cycles
- Total: Total of all reporting groups
Arm/Group | TAC X 6 | AC X 4 Then P X 4 | AC X 4 Then PG X 4 | Total
Number analyzed (Participants) | 1623 | 1623 | 1621 | 4867
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9.5) | 51 (9.5) | 51 (9.4) | 51 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1623 | 1623 | 1621 | 4867
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival: Any Recurrence, Contralateral Breast Cancer, Second Primary Cancer, Death From Any Cause Prior to Recurrence or Second Primary Cancer
Description: The percentage of patients alive and cancer-free.
Time Frame: 5 years
Population: For Arm 1 there is no follow-up data for 20 participants; for Arm 2 there is no follow-up data for 16 participants; and for Arm 3 there is no follow-up data for 17 participants.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Group 1: TAC X 6 | Group 2: AC X 4 Then P X 4 | Group 3: AC X 4 Then PG X 4
Number analyzed (Participants) | 1610 | 1618 | 1613
percentage of patients | 80.1 [78.0 to 82.0] | 82.2 [80.2 to 84.0] | 80.6 [78.5 to 82.5]

2. Secondary Outcome: Overall Survival
Description: Percentage of participants alive at 5 years
Time Frame: 5 years
Population: For Arm 1 there is no follow-up data for 13 participants; for Arm 2 there is no follow-up data for 10 participants; and for Arm 3 there is no follow-up data for 12 participants.
Measure: Number (95% Confidence Interval); unit: percentage of patients alive
Arm/Group | Group 1: TAC X 6 | Group 2: AC X 4 Then P X 4 | Group 3: AC X 4 Then PG X 4
Number analyzed (Participants) | 1617 | 1624 | 1618
percentage of patients alive | 89.6 [88.1 to 91.1] | 89.1 [87.4 to 90.5] | 90.8 [89.3 to 92.1]

3. Secondary Outcome: Recurrence-free Interval: Time to First Local, Regional, or Distant Recurrence
Description: Percentage of patients recurrence-free (no first local, regional, or distant recurrence)
Time Frame: 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Group 1: TAC X 6 | Group 2: AC X 4 Then P X 4 | Group 3: AC X 4 Then PG X 4
Number analyzed (Participants) | 1610 | 1618 | 1613
percentage of patients | 85.1 [83.2 to 86.9] | 86.2 [84.3 to 87.9] | 84.8 [82.8 to 86.5]

4. Secondary Outcome: Distant Recurrence-free Interval: the Time to Distant Disease Recurrence Only
Description: Percentage of patients distant recurrence-free (no distant disease recurrence only)
Time Frame: 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Group 1: TAC X 6 | Group 2: AC X 4 Then P X 4 | Group 3: AC X 4 Then PG X 4
Number analyzed (Participants) | 1610 | 1618 | 1613
percentage of patients | 86.6 [84.7 to 88.2] | 87.4 [85.6 to 89.0] | 86.6 [84.7 to 88.2]

5. Secondary Outcome: Toxicity
Description: Percentage of patients who ever experienced grade 2 or higher toxicities.
Time Frame: 30 days after the last dose of study therapy (about 7 months after study entry)
Population: For Arm 1 there is no follow-up data for 23 participants; for Arm 2 there is no follow-up data for 11 participants; and for Arm 3 there is not follow-up data for 18 participants.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Group 1: TAC X 6 | Group 2: AC X 4 Then P X 4 | Group 3: AC X 4 Then PG X 4
Number analyzed (Participants) | 1607 | 1623 | 1612
percentage of patients | 82.7 [80.8 to 84.5] | 87.5 [85.8 to 89.0] | 88.4 [86.7 to 89.9]

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Groups:
- TAC X 6: TAC X 6
- AC X 4 Then P X 4: AC X 4 then P X 4
- AC X 4 Then PG X 4: AC X 4 then PG X 4
Arm/Group | TAC X 6 | AC X 4 Then P X 4 | AC X 4 Then PG X 4
Serious Adverse Events (participants affected / at risk) | 277/1601 | 158/1612 | 187/1604
Other Adverse Events (participants affected / at risk) | 1231/1601 | 1322/1612 | 1323/1604
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAC X 6 (N=1601) | AC X 4 Then P X 4 (N=1612) | AC X 4 Then PG X 4 (N=1604)
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 21 | 8 | 13
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4
Alanine aminotransferase increased (ALT/SGPT) (Investigations) | 4 | 7 | 5
Anorexia (Metabolism and nutrition disorders) | 3 | 3 | 4
Anxiety (Psychiatric disorders) | 3 | 1 | 2
Aspartate aminotransferase increased (AST/SGOT) (Investigations) | 5 | 6 | 4
Atrial fibrillation (Cardiac disorders) | 2 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bladder infection (Infections and infestations) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 12 | 9
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Cardiac troponin I increased (Investigations) | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 9 | 2 | 2
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 2 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 3
Creatinine increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 22 | 42 | 23
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 4 | 2 | 4
Diarrhea (Gastrointestinal disorders) | 9 | 17 | 47
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 | 23 | 14
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Esophageal ulcer (Gastrointestinal disorders) | 2 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 3 | 1 | 0
Fatigue (General disorders) | 43 | 37 | 27
Febrile neutropenia (Blood and lymphatic system disorders) | 40 | 45 | 132
Fever (General disorders) | 3 | 10 | 3
Flushing (Vascular disorders) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 4 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 6
Hematoma (Vascular disorders) | 2 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 2 | 0
Hot flashes (Vascular disorders) | 1 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 2 | 5 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 10
Ileus (Gastrointestinal disorders) | 1 | 1 | 0
Injection site reaction (General disorders) | 1 | 0 | 0
INR increased (Investigations) | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0
Ischemia cerebrovascular (Nervous system disorders) | 1 | 2 | 0
Lipase increased (Investigations) | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 2 | 3
Mucositis oral (Gastrointestinal disorders) | 3 | 4 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 9 | 10
Nausea (Gastrointestinal disorders) | 26 | 35 | 18
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 20 | 5 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 8 | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 2 | 9
Platelet count decreased (Investigations) | 3 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 16 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Psychosis (Psychiatric disorders) | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 2 | 1 | 0
Seizure (Nervous system disorders) | 3 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 1 | 0
Syncope (Nervous system disorders) | 10 | 6 | 8
Typhlitis (Gastrointestinal disorders) | 3 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 22 | 14 | 23
Weight loss (Investigations) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 1 | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 3 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 1 | 3
Localized edema (General disorders) | 1 | 0 | 0
Gallbladder infection (Infections and infestations) | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAC X 6 (N=1601) | AC X 4 Then P X 4 (N=1612) | AC X 4 Then PG X 4 (N=1604)
Abdominal pain (Gastrointestinal disorders) | 93 | 67 | 87
Alanine aminotransferase increased (ALT/SGPT) (Investigations) | 27 | 73 | 108
Bone pain (Musculoskeletal and connective tissue disorders) | 267 | 484 | 446
Constipation (Gastrointestinal disorders) | 154 | 204 | 184
Cough (Respiratory, thoracic and mediastinal disorders) | 64 | 82 | 83
Dehydration (Metabolism and nutrition disorders) | 137 | 87 | 94
Diarrhea (Gastrointestinal disorders) | 325 | 159 | 185
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 110 | 136 | 124
Fatigue (General disorders) | 805 | 784 | 774
Febrile neutropenia (Blood and lymphatic system disorders) | 144 | 50 | 50
Fever (General disorders) | 91 | 63 | 69
Headache (Nervous system disorders) | 142 | 182 | 188
Mucositis oral (Gastrointestinal disorders) | 173 | 157 | 201
Myalgia (Musculoskeletal and connective tissue disorders) | 256 | 536 | 512
Nausea (Gastrointestinal disorders) | 510 | 504 | 497
Peripheral motor neuropathy (Nervous system disorders) | 37 | 86 | 76
Peripheral sensory neuropathy (Nervous system disorders) | 167 | 484 | 428
Vomiting (Gastrointestinal disorders) | 284 | 245 | 306

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days